CLINICAL TRIAL: NCT03435588
Title: Endoscopic Ultrasound (EUS)-Guided Fine Needle Aspiration (FNA) With Rapid On-site Evaluation (ROSE) of Cytopathology vs. EUS-guided Fine Needle Biopsy (FNB) Alone in the Diagnosis of Pancreatic Solid Lesions: a Randomized Controlled Trial
Brief Title: Endoscopic Ultrasound (EUS)-Guided Fine Needle Aspiration (FNA) With Rapid On-site Evaluation (ROSE) of Cytopathology vs. EUS-guided Fine Needle Biopsy (FNB) Alone in the Diagnosis of Pancreatic Solid Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Yen-I Chen, Assistant Professor of Medicine, Division of Gastroenterology and Hepatology, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 22125
Record Dates: First submitted 2018-01-15; First posted 2018-02-19 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Solid Pancreatic Tumor

STUDY DESIGN:
Intervention Model Description: Procedures are performed with a linear echoendoscope under conscious sedation. EUS-FNB is performed with a 22G or 25G needles Core-needle. Tissue sampling technique is standardized between the endoscopists. Two passes are performed using the core needle. A third pass is allowed if, on macroscopic inspection of the acquired sample, the specimen is deemed insufficient by the endoscopist. EUS-FNA with ROSE is performed with a 22 or 25 gauge FNA needle.
  This is a multi-center, randomized, single blinded, non-inferiority, trial comparing EUS-FNB alone to EUS-FNA with ROSE in the diagnosis of solid pancreatic masses. Following consent, patients are randomized, at the time of the procedure, to undergo either EUS-FNB alone or EUS-FNA with ROSE. The randomization sequence will be generated by a computerized randomization scheme using a block size of 10 stratified according to the endoscopist.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-FNA with ROSE (Active Comparator): EUS-FNA with ROSE is performed with a 22 or 25 gauge FNA needle. The sampled specimen is expressed into a glass slide with a stylet; then using another glass slide the sample is spread out to make smears on two slides. Each pair of slides is then numbered according to their respective needle passes. One slide is air dried and stained with modified Giemsa stain for ROSE, while the other slide is fixed in 95% ethanol and later coated with with Papanicolaou stain.
  Interventions: Procedure: EUS; Procedure: FNA with ROSE
- EUS-FNB alone (Experimental): EUS-FNB is performed with a 22 or 25 gauge Core-needle. Tissue sampling technique is standardized between the endoscopists. Two passes are performed using the core needle. The biopsied samples are then expressed using a stylet into a jar filled with 10% formalin. A third pass is allowed if, on macroscopic inspection of the acquired sample, the specimen is deemed insufficient by the endoscopist.
  Interventions: Procedure: EUS; Procedure: FNB alone

INTERVENTIONS:
Procedure: EUS — Radial endoscopic ultrasound. A special endoscope uses high-frequency sound waves to produce detailed images of the lining and walls of the digestive tract , and allows to take samples from abnormal areas.
Procedure: FNA with ROSE — Endoscopic ultrasound guided biopsy of the pancreas with the traditional fine needle aspirate needle with the addition of rapid on-site cytopathology (cytopathologist looking at each biopsy samples as they are taken): The sampling is done with a small needle called fine needle aspiration needle or FNA. FNA alone is sometimes limited due to inadequate acquisition of cells for proper diagnosis under the microscope, which can lead to need for repeat endoscopic procedures and delay in diagnosis and possibly treatment. Rapid on-site evaluation of cytopathology (ROSE) is where a cytopathologist is next to the physician doing the endoscopic procedures and evaluates each sampling performed.
  Arms: EUS-FNA with ROSE
Procedure: FNB alone — Endoscopic ultrasound guided biopsy with a novel core biopsy needle without on-site cytopathology: New needles called core needles (fine needle biopsy, FNB) have recently been developed which not only acquires cells but also the entire tissue structure (histology).
  Arms: EUS-FNB alone

SUMMARY:
Currently, the best way to evaluate pancreatic masses is through endoscopic-guided needle sampling of the mass to determine the diagnosis by looking at the acquired tissue under a microscope. This is done by inserting a small camera (endoscope) through the mouth of the patient then advanced to the stomach and using ultrasound guidance a sample of the pancreas can be acquired through the stomach. The sampling is usually done with a small needle called fine needle aspiration needle or FNA. FNA alone is sometimes limited due to inadequate acquisition of cells for proper diagnosis under the microscope, which can lead to need for repeat endoscopic procedures and delay in diagnosis and possibly treatment. Rapid on-site evaluation of cytopathology (ROSE) is where a cytopathologist is next to the physician doing the endoscopic procedures and evaluates each sampling performed immediately under the microscope and can give feedback to the endoscopist until enough cells has been acquired for a diagnosis. This method has been shown to increase the ability to diagnose pancreatic cancer but is expensive and requires significant amount of resources. New needles called core needles (fine needle biopsy, FNB) have recently been developed which not only acquires cells but also the entire tissue structure (histology) and has been shown to be also very accurate in the diagnosis of pancreatic cancer.

The purpose of this study is to compare endoscopy-guided biopsy of pancreatic masses with the new core needle (FNB), which can obtain more tissue for diagnosis vs. using a traditional needle (FNA) with the help of an immediate assessment of the obtained samples under the microscope to determine whether enough tissue has been obtained (ROSE). Both approaches have been shown to increase the accuracy of diagnosis in solid pancreatic masses but it is unclear which one is superior. This is a randomized trial meaning that the participants would either undergo biopsy with the new needle or with the traditional needle plus the addition of on-site assessment of the obtained samples. The advantage of the new needle is that it is easy to implement and likely much cheaper. If the investigators can show in our study that the new needles are as accurate as FNA with ROSE then FNB could be implemented across hospitals worldwide in an easier and less expensive fashion.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients referred for EUS evaluation of a definite solid pancreatic mass noted on computed tomography(CT)/Magnetic resonance imaging(MRI)/EUS, in which malignancy is suspected with no previous histological diagnosis

Exclusion Criteria:

* Age < 18 years, pregnant patients.
* Uncorrectable coagulopathy Prothrombin time (PT) >50% of control, Partial Thromboplastin time (PTT) >50 sec, or International normalized ratio (INR) >1.5 and/or uncorrectable thrombocytopenia platelet count<50, 000109/L.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 12 months
  Defined as (true positive + true negative)/all samples
Final diagnosis of malignant pancreatic mass | 10 months
  Will be based on the following criteria:
  * Histological evidence of malignancy on the corresponding subsequent surgical specimen
  * Presence of an unresectable lesion during subsequent surgery
  * Malignant cytology/pathology on EUS-sampling followed by documented loco-regional progression/development of metastases on follow-up axial imaging.
Final diagnosis of benign pancreatic mass | 10 months
  Will be based on the following criteria:
  * Surgical pathology or exploration showing the absence of malignancy
  * Follow-up imaging at > 6 months reporting stability of the pancreatic lesion
  * Cytological or histopathological diagnosis of benign disease with an appropriate clinical course of disease for minimum of 6 months

SECONDARY OUTCOMES:
Diagnostic characteristics | 6 to 12 months of data collection and 3 to 6 months of data analysis.
  sensitivity, specificity, positive and negative predictive value
Specimen adequacy | 6 to 12 months of data collection and 3 to 6 months of data analysis.
  Defined as the proportion of samples in which a final histopathological diagnosis could be made
Median number of needle passes | 6 to 12 months of data collection and 3 to 6 months of data analysis.
  Number of times passing the needle for tissue acquisition
Procedural time | 6 to 12 months of data collection and 3 to 6 months of data analysis.
  Time spent during the procedure
Rate of procedure-related adverse events | 6 to 12 months of data collection and 3 to 6 months of data analysis.
  An adverse event is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a procedure done, whether or not considered causally related to the procedure.
  A serious adverse event is an adverse event occurring during the procedure or any time after the procedure, that fulfills one or more of the following criteria:
  * Results in death
  * Is immediately life-threatening
  * Requires in-patient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability or incapacity
  * Is a congenital abnormality or birth defect
  * Is an important medical event that may jeopardize the patient or may require medical intervention to prevent one of the outcomes listed above.

CONTACTS AND LOCATIONS:
Overall Officials: Yen-I Chen, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (6):
- Canada (6):
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Moncton Hospital, Moncton, New Brunswick
  - The Ottawa Hospital, Ottawa, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

REFERENCES:
- [Background] Klapman JB, Logrono R, Dye CE, Waxman I. Clinical impact of on-site cytopathology interpretation on endoscopic ultrasound-guided fine needle aspiration. Am J Gastroenterol. 2003 Jun;98(6):1289-94. doi: 10.1111/j.1572-0241.2003.07472.x. PMID 12818271
- [Background] Gress FG, Hawes RH, Savides TJ, Ikenberry SO, Lehman GA. Endoscopic ultrasound-guided fine-needle aspiration biopsy using linear array and radial scanning endosonography. Gastrointest Endosc. 1997 Mar;45(3):243-50. doi: 10.1016/s0016-5107(97)70266-9. PMID 9087830
- [Background] Chang KJ, Katz KD, Durbin TE, Erickson RA, Butler JA, Lin F, Wuerker RB. Endoscopic ultrasound-guided fine-needle aspiration. Gastrointest Endosc. 1994 Nov-Dec;40(6):694-9. PMID 7859967
- [Background] Kulesza P, Eltoum IA. Endoscopic ultrasound-guided fine-needle aspiration: sampling, pitfalls, and quality management. Clin Gastroenterol Hepatol. 2007 Nov;5(11):1248-54. doi: 10.1016/j.cgh.2007.09.011. PMID 17981244
- [Background] Kandel P, Tranesh G, Nassar A, Bingham R, Raimondo M, Woodward TA, Gomez V, Wallace MB. EUS-guided fine needle biopsy sampling using a novel fork-tip needle: a case-control study. Gastrointest Endosc. 2016 Dec;84(6):1034-1039. doi: 10.1016/j.gie.2016.03.1405. Epub 2016 Mar 24. PMID 27018087
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503
- [Derived] Chen YI, Chatterjee A, Berger R, Kanber Y, Wyse J, Lam E, Gan I, Auger M, Kenshil S, Telford J, Donnellan F, Quinlan J, Lutzak G, Alshamsi F, Parent J, Waschke K, Alghamdi A, Barkun J, Metrakos P, Chaudhury P, Martel M, Dorreen A, Candido K, Miller C, Adam V, Barkun A, Zogopoulos G, Wong C. Endoscopic ultrasound (EUS)-guided fine needle biopsy alone vs. EUS-guided fine needle aspiration with rapid onsite evaluation in pancreatic lesions: a multicenter randomized trial. Endoscopy. 2022 Jan;54(1):4-12. doi: 10.1055/a-1375-9775. Epub 2021 Apr 15. PMID 33506455

DOCUMENTS (2):
  • Informed Consent Form (2018-02-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT03435588/ICF_000.pdf
  • Study Protocol (2018-02-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT03435588/Prot_001.pdf